CLINICAL TRIAL: NCT06551129
Title: Real-World Camzyos Patient Reported OutcoMes Through PAtient SurveyS in Hypertrophic CardioMyopathy (COMPASS-HCM): A Prospective Longitudinal Study
Brief Title: Real-world Patient Reported Outcomes Among Patients Treated With Camzyos
Acronym: COMPASS-HCM
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV027-1002
Record Dates: First submitted 2024-08-06; First posted 2024-08-13 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy
Keywords: Obstructive Hypertrophic cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mavacamten: Adult participants with symptomatic obstructive hypertrophic cardiomyopathy treated with mavacamten
  Interventions: Drug: Mavacamten

INTERVENTIONS:
Drug: Mavacamten — As prescribed by treating physician

SUMMARY:
This real-world study will assess changes in health status among participants with symptomatic obstructive hypertrophic cardiomyopathy who are treated with mavacamten in the real world.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥18 years of age.
* Participants who are prescribed mavacamten for obstructive hypertrophic cardiomyopathy
* Provided informed consent to participate in the study

Exclusion Criteria:

* Previously or currently enrolled in clinical trials for any cardiac myosin inhibitors
* Treated for >7 days with mavacamten by the day of completing the baseline survey
* Enrolled in any clinical trials at the time of or within the six-month period prior to the screening
* Had heart attack requiring coronary artery bypass grafting within the three-month period prior to the screening
* Had stroke or transient ischemic attack within the six-month period prior to the screening
* Had moderate-to-severe lung disease which impacted the ability to perform daily activities of living and ability to breathe
* Had major lung (thoracic) or heart (cardiac) surgery within the six-month period prior to the screening
* Scheduled for a major surgery for the next three months, such as joint surgeries including hip replacement, abdominal surgeries, lung surgeries, heart surgeries, eye surgeries, brain surgeries, and any other major surgeries that require general anesthesia and at least an overnight hospital stay
* Hospitalized requiring an overnight stay at the time of or within the two-week period prior to the screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants in the United States diagnosed with obstructive hypertrophic cardiomyopathy (oHCM) receiving mavacamten treatment
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Participant Hypertrophic Cardiomyopathy symptoms as assessed by Hypertrophic Cardiomyopathy Symptom Questionnaire (HCMSQ v2,0 - 7-day recall version) | Baseline and weeks 2, 4, 8, 12, 24, 30, 48, 60, 72, 84 and 96
Participant physical limitation, symptom stability, symptom frequency, symptom burden, self-efficacy, QoL, and social limitations as assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ-23) | Baseline and weeks 2, 4, 8, 12, 24, 30, 48, 60, 72, 84 and 96
Participant mavacamten treatment status | Weeks 2, 4, 8, 12, 24, 30, 48, 60, 72, 84 and 96
Other pharmacological and surgical treatments for obstructive hypertrophic cardiomyopathy (HCM) | Baseline and weeks 2, 4, 8, 12, 24, 30, 48, 60, 72, 84 and 96
Participant symptom severity as assessed by self-assessed New York Heart Association (SA-NYHA) functional class | Baseline and weeks 2, 4, 8, 12, 24, 30, 48, 60, 72, 84 and 96
Participant change in symptom severity as assessed by Patient Global Impression of Change (PGI-C) | Weeks 2, 4, 8, 12, 24, 30, 48, 72, and 96
Participant septal reduction therapy | Baseline and weeks 12, 30, 48 and 96
Participant major injury or surgery since previous survey | Weeks 2, 4, 8, 12, 24, 30, 48, 60, 72, 84 and 96
Participant survey response on experience with CAMZYOS Risk Evaluation and Mitigation Strategy program (REMS) Program | Baseline and weeks 4, 12, 30, 48, 72 and 96
Participant medical history | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Analysis Group Inc., Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts